CLINICAL TRIAL: NCT03253393
Title: Microbial Contamination Rates on the Back Surface of Soft Contact Lenses in Two Short-term, Randomized, Contralateral Non-dispensing Studies
Brief Title: Smart Touch Non-dispensing Handling Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Collaborators: Menicon Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jacqueline Tan-Showyin, Senior Research Fellow, The University of New South Wales
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SOVS2017-050
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Results first posted 2021-11-02 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Optometry

STUDY DESIGN:
Intervention Model Description: Contralateral study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Silicone hydrogel (with EDTA) in Smart Touch vs. in conventional packaging (Experimental): Silicone hydrogel (with EDTA) in Smart Touch vs. in conventional packaging
  Interventions: Device: Smart Touch Technology packaging; Device: Conventional lens packaging
- Hydrogel (no EDTA) in Smart Touch vs. in conventional packaging (Experimental): Hydrogel (no EDTA) in Smart Touch vs. in conventional packaging
  Interventions: Device: Smart Touch Technology packaging; Device: Conventional lens packaging
- Silicone hydrogel (no EDTA) vs. hydrogel (with EDTA) in Smart Touch (Experimental): Silicone hydrogel (no EDTA) vs. hydrogel (with EDTA) in Smart Touch
  Interventions: Device: EDTA

INTERVENTIONS:
Device: Smart Touch Technology packaging — hioxifilcon A contact lens in Smart Touch Technology (hydrogel, no EDTA) midafilcon A contact lens in Smart Touch Technology (silicone hydrogel, with EDTA)
  Arms: Hydrogel (no EDTA) in Smart Touch vs. in conventional packaging; Silicone hydrogel (with EDTA) in Smart Touch vs. in conventional packaging
Device: Conventional lens packaging — hioxifilcon A contact lens in conventional lens packaging (hydrogel, no EDTA) midafilcon A contact lens in conventional lens packaging (silicone hydrogel, with EDTA)
  Arms: Hydrogel (no EDTA) in Smart Touch vs. in conventional packaging; Silicone hydrogel (with EDTA) in Smart Touch vs. in conventional packaging
Device: EDTA — hioxifilcon A contact lens in Smart Touch Technology (hydrogel, with EDTA) midafilcon A contact lens in Smart Touch Technology (silicone hydrogel, no EDTA)
  Arms: Silicone hydrogel (no EDTA) vs. hydrogel (with EDTA) in Smart Touch

SUMMARY:
This study is a randomized, contralateral, investigator-masked non-dispensing study, to investigate the microbial contamination rates on the back surface of two types of soft contact lenses (hydrogel and silicone hydrogel) extracted from Smart Touch Technology blister packs versus conventional lens packaging after short-term placement on the eye, and to compare the microbial contamination rates of the worn contact lenses to those on the participants' hands/fingers used to conduct lens insertion.

DETAILED DESCRIPTION:
This will be a prospective, single centre, randomized, contralateral, investigator-masked non-dispensing study. This study requires three visits of approx. 1 hour duration each.

At the first visit, the order in which the hydrogel (no EDTA) and silicone hydrogel (with EDTA) contact lenses are allocated to the study participants will be randomized. At the second visit, participants will be crossed over to the alternate lens type (hydrogel no EDTA or silicone hydrogel with EDTA).

At the third visit, participants will be randomly allocated to wear the hydrogel lens (with EDTA) in one eye and the silicone hydrogel lens (no EDTA) in the other eye, both removed from Smart Touch Technology packaging.

At each visit, participants will be instructed to:

* Wash their hands prior to handling the contact lenses;
* Swab their thumb and two index fingers of the hand routinely used to conduct contact lens insertion using a sterile cotton swab moistened with sterile preservative free saline for the evaluation of skin microbiota;
* Follow the manufacturer's guidelines for lens insertion;
* Open the blister pack and insert the contact lens randomly assigned for the right eye;
* Open the blister pack and insert the contact lens assigned for the left eye;
* Contact lenses will be removed aseptically by a masked investigator after 45 minutes of lens wear.

Lenses and finger swabs will be analysed for microbial contamination using established routine microbiology protocols. The number and species of organisms will be determined.

A minimum washout period of 48 hours will occur between the study visits.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and comprehend English and give informed consent as demonstrated by signing a Participant Information Statement and Consent Form;
* Be at least 18 years old;
* Experienced soft contact lens wearer;
* Willing to refrain from wearing contact lenses for 24 hours prior to the scheduled study visit

Exclusion Criteria:

* Under 18 years old;
* Have any active corneal infection, ocular disease or systemic disease that would affect wearing of contact lenses;
* Use or have a need for any systemic or topical medications which may alter normal ocular findings/are known to affect a participant's ocular health/physiology either in an adverse manner or risk providing a false positive;
* Have had eye surgery within 12 weeks immediately prior to enrolment for this trial;
* Have contraindications to contact lens wear;
* Have a greater than 2 line reduction in habitual visual acuity while wearing the study contact lenses;
* Be currently enrolled in another clinical trial;
* Be pregnant (verbal self-report)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Optometry and Vision Science, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tan J, Siddireddy JS, Wong K, Shen Q, Vijay AK, Stapleton F. Factors Affecting Microbial Contamination on the Back Surface of Worn Soft Contact Lenses. Optom Vis Sci. 2021 May 1;98(5):512-517. doi: 10.1097/OPX.0000000000001693. PMID 33973914

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25 subjects were required to complete each of the three study interventions
Pre-assignment Details: 25 subjects were enrolled and randomised. Of those randomised, 13 did not complete the third visit/intervention. Therefore an additional 13 subjects were recruited to complete the third intervention only.
Groups:
- SiH (With EDTA) , Then H (no EDTA), Then SiH (Without EDTA) and H (With EDTA) in Smart Touch: Participants first received a Silicone Hydrogel lens (with EDTA) in Smart Touch packaging which was inserted in one eye and a Silicone Hydrogel lens (with EDTA) in a conventional blister which was inserted in the other eye. After a minimum washout period of 48 hours, they then received a Hydrogel lens (no EDTA) in Smart Touch packaging which was inserted in one eye and a Hydrogel lens in a conventional blister which was inserted in the other eye. After a minimum washout period of 48 hours they then received a Silicone Hydrogel lens (without EDTA) in Smart Touch packaging in one eye and a Hydrogel lens (with EDTA) in Smart Touch packaging in the other eye.
  Smart Touch Technology packaging: midafilcon A contact lens in Smart Touch Technology Flat Pack (silicone hydrogel, with EDTA)
  Conventional lens packaging: hioxifilcon A contact lens in conventional lens packaging (hydrogel, no EDTA) asmofilcon A contact lens in conventional lens packaging (silicone hydrogel, with EDTA)
- H (no EDTA), Then SiH (With EDTA), Then SiH (Without EDTA) vs H (With EDTA) in Smart Touch: Participants first received a Hydrogel lens (no EDTA) in Smart Touch packaging which was inserted in one eye and a Hydrogel lens in a conventional blister which was inserted in the other eye. After a minimum washout period of 48 hours, they then received a Silicone Hydrogel lens (with EDTA) in Smart Touch packaging which was inserted in one eye and a Silicone Hydrogel lens (with EDTA) in a conventional blister which was inserted in the other eye. After a minimum washout period of 48 hours they then received a Silicone Hydrogel lens (without EDTA) in Smart Touch packaging in one eye and a Hydrogel lens (with EDTA) in Smart Touch packaging in the other eye.
- SiH (Without EDTA) in Smart Touch vs H (With EDTA) in Smart Touch: Participants received a Silicone Hydrogel lens (without EDTA) in Smart Touch packaging which was inserted in one eye and a Hydrogel lens (with EDTA) in Smart Touch packaging which was inserted in the other eye.
Period: First Intervention
Arm/Group | SiH (With EDTA) , Then H (no EDTA), Then SiH (Without EDTA) and H (With EDTA) in Smart Touch | H (no EDTA), Then SiH (With EDTA), Then SiH (Without EDTA) vs H (With EDTA) in Smart Touch | SiH (Without EDTA) in Smart Touch vs H (With EDTA) in Smart Touch
Started | 12 | 13 | 0
Completed | 12 | 13 | 0
Not Completed | 0 | 0 | 0
Period: Washout (Minimum 48 Hours)
Arm/Group | SiH (With EDTA) , Then H (no EDTA), Then SiH (Without EDTA) and H (With EDTA) in Smart Touch | H (no EDTA), Then SiH (With EDTA), Then SiH (Without EDTA) vs H (With EDTA) in Smart Touch | SiH (Without EDTA) in Smart Touch vs H (With EDTA) in Smart Touch
Started | 12 | 13 | 0 (Participants in this group were only assigned to one visit/intervention)
Completed | 12 | 13 | 0 (Participants in this group were only assigned to one visit/intervention)
Not Completed | 0 | 0 | 0
Period: Second Intervention
Arm/Group | SiH (With EDTA) , Then H (no EDTA), Then SiH (Without EDTA) and H (With EDTA) in Smart Touch | H (no EDTA), Then SiH (With EDTA), Then SiH (Without EDTA) vs H (With EDTA) in Smart Touch | SiH (Without EDTA) in Smart Touch vs H (With EDTA) in Smart Touch
Started | 12 | 13 | 0 (Participants in this group were only assigned to one visit/intervention)
Completed | 12 | 13 | 0 (Participants in this group were only assigned to one visit/intervention)
Not Completed | 0 | 0 | 0
Period: Washout (Minimum 48 Hours)
Arm/Group | SiH (With EDTA) , Then H (no EDTA), Then SiH (Without EDTA) and H (With EDTA) in Smart Touch | H (no EDTA), Then SiH (With EDTA), Then SiH (Without EDTA) vs H (With EDTA) in Smart Touch | SiH (Without EDTA) in Smart Touch vs H (With EDTA) in Smart Touch
Started | 12 | 13 | 0 (Participants in this group were only assigned to one visit/intervention)
Completed | 6 | 6 | 0 (Participants in this group were only assigned to one visit/intervention)
Not Completed | 6 | 7 | 0
Not completed — 13 participants exited study after first two visits/interventions | 6 | 7 | 0
Period: Third Intervention
Arm/Group | SiH (With EDTA) , Then H (no EDTA), Then SiH (Without EDTA) and H (With EDTA) in Smart Touch | H (no EDTA), Then SiH (With EDTA), Then SiH (Without EDTA) vs H (With EDTA) in Smart Touch | SiH (Without EDTA) in Smart Touch vs H (With EDTA) in Smart Touch
Started | 6 | 6 | 13 (Participants in this group were only assigned to one visit/intervention)
Completed | 6 | 6 | 13 (Participants in this group were only assigned to one visit/intervention)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SiH (With EDTA) , Then H (no EDTA), Then SiH (Without EDTA) and H (With EDTA) in Smart Touch: Participants first received a Silicone Hydrogel lens (with EDTA) in Smart Touch packaging which was inserted in one eye and a Silicone Hydrogel lens (with EDTA) in a conventional blister which was inserted in the other eye. After a minimum washout period of 48 hours, they then received a Hydrogel lens (no EDTA) in Smart Touch packaging which was inserted in one eye and a Hydrogel lens in a conventional blister which was inserted in the other eye. After a minimum washout period of 48 hours they then received a Silicone Hydrogel lens (without EDTA) in Smart Touch packaging in one eye and a Hydrogel lens (with EDTA) in Smart Touch packaging in the other eye.
- Total: Total of all reporting groups
Arm/Group | SiH (With EDTA) , Then H (no EDTA), Then SiH (Without EDTA) and H (With EDTA) in Smart Touch | H (no EDTA), Then SiH (With EDTA), Then SiH (Without EDTA) vs H (With EDTA) in Smart Touch | SiH (Without EDTA) in Smart Touch vs H (With EDTA) in Smart Touch | Total
Number analyzed (Participants) | 12 | 13 | 13 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 1
  Between 18 and 65 years | 12 | 13 | 10 | 35
  >=65 years | 0 | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (8.8) | 29.8 (8.8) | 30.1 (14.2) | 29.9 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 9 | 24
  Male | 5 | 5 | 4 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8 | 10 | 8 | 26
  Non-Asian | 4 | 3 | 5 | 12
Region of Enrollment [Number; unit: participants]
  Australia | 12 | 13 | 13 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Without Contamination of Contact Lenses
Description: Number of Participants Without Contamination of Contact Lenses after 45 minutes of wear
Time Frame: After 45 minutes of lens wear
Measure: Count of Participants; unit: Participants
Groups:
- Silicone Hydrogel (With EDTA) in Smart Touch: Lens Contamination for Silicone Hydrogel lenses in Smart Touch™ (with EDTA).
- Silicone Hydrogel (With EDTA) in Conventional Packaging: Lens Contamination for Silicone hydrogel (with EDTA) in conventional packaging
- Silicone Hydrogel (no EDTA) in Smart Touch: Lens Contamination for Silicone Hydrogel lenses in Smart Touch™ (no EDTA).
- Hydrogel (no EDTA) in Smart Touch: Lens Contamination for Hydrogel lenses in Smart Touch™ (no EDTA).
- Hydrogel (no EDTA) in Conventional Packaging: Lens Contamination for Hydrogel in Conventional packaging (no EDTA).
- Hydrogel (With EDTA) in Smart Touch: Lens Contamination for Hydrogel lenses in Smart Touch™ (with EDTA).
Arm/Group | Silicone Hydrogel (With EDTA) in Smart Touch | Silicone Hydrogel (With EDTA) in Conventional Packaging | Silicone Hydrogel (no EDTA) in Smart Touch | Hydrogel (no EDTA) in Smart Touch | Hydrogel (no EDTA) in Conventional Packaging | Hydrogel (With EDTA) in Smart Touch
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25
Participants | 16 | 9 | 4 | 14 | 7 | 16

2. Secondary Outcome: Bacterial Counts of Worn Contact Lenses
Description: Bacterial counts of contact lenses after 45 minutes of wear (CFU count /lens)
Time Frame: After 45 minutes of lens wear
Measure: Median (Inter-Quartile Range); unit: CFU count per lens
Units Other Than Participants: Lens
Arm/Group | Silicone Hydrogel (With EDTA) in Smart Touch | Silicone Hydrogel (With EDTA) in Conventional Packaging | Silicone Hydrogel (no EDTA) in Smart Touch | Hydrogel (no EDTA) in Smart Touch | Hydrogel (no EDTA) in Conventional Packaging | Hydrogel (With EDTA) in Smart Touch
Number analyzed (Participants) | 25 | 25 | 25 | 25 | 25 | 25
Number analyzed (Lens) | 25 | 25 | 25 | 25 | 25 | 25
CFU count per lens | 0 [0 to 43] | 1 [0 to 25] | 4 [0 to 10] | 0 [0 to 17] | 1 [0 to 16] | 0 [0 to 9]

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events occurring during lens wear i.e. 45 minutes for each visit, up to 3 visits.
Description: Participants were monitored for adverse events at each visit
Arm/Group | Silicone Hydrogel (With EDTA) in Smart Touch | Silicone Hydrogel (With EDTA) in Conventional Packaging | Silicone Hydrogel (no EDTA) in Smart Touch | Hydrogel (no EDTA) in Smart Touch | Hydrogel (no EDTA) in Conventional Packaging | Hydrogel (With EDTA) in Smart Touch
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT03253393/Prot_SAP_000.pdf